CLINICAL TRIAL: NCT00194545
Title: Effect of Medication Diaries on Adherence to Highly Active Antiretroviral Drugs Among HIV-1 Infected Kenyan Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-1519-D 02
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: HIV Infections
Keywords: HIV-1; pediatric adherence; medication diaries; HAART; Treatment Naive
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Medication diary
  Interventions: Behavioral: Medication diaries
- 2 (No Intervention): Caregivers only receive counseling which is the standard of care

INTERVENTIONS:
Behavioral: Medication diaries — Caregivers expected to complete medication diaries daily
  Arms: 1

SUMMARY:
Following significant reduction in antiretroviral drug prices over the past two years, more HIV-1 infected African adults and children are gaining access to treatment. However, due to complex drug regimens that have to be taken continuously, suboptimal adherence is likely to be a formidable challenge. As programs providing antiretroviral drugs in Africa scale up, achievement of excellent adherence is a high priority as this will result in maximum benefits from the drugs and forestall development of resistant virus. A better understanding of predictors of pediatric HAART adherence in African children is essential in order to formulate feasible, culturally appropriate, strategies to monitor and enhance adherence. There is also urgent need to evaluate simple, inexpensive interventions that are widely applicable in the African setting. The medication diary has been used empirically among HIV infected adults and children in Western countries, mainly as a tool for monitoring and to a lesser extent improving HAART adherence. Literacy levels have risen significantly in most African regions over the past few years, and the diary can also be further modified using pictures to suit parents of different literacy levels. We propose to conduct a randomized control trial to determine the effect of medication diaries and counseling versus counseling alone on HAART-adherence in HIV-1 infected children and their parents/caregivers in Nairobi Kenya.

DETAILED DESCRIPTION:
Study design: This is a randomized trial comparing adherence to antiretroviral drugs and clinical outcomes between 50 HIV-1 infected Kenyan children randomized to a simple medication diary plus standard counseling with a similar group of children randomized to counseling alone.

Study procedures:

Parents or caregivers of HIV-1 infected children discharged from the Kenyatta National Hospital (KNH) children's wards or seen in pediatric outpatient clinics will be invited to participate in the study by nurse counselors. Informed written consent will be obtained from those who meet eligibility criteria and agree to participate. The consenting process will be done by the principal investigator in a confidential area. A baseline questionnaire will be administered to obtain socio-demographic information and previous medical history of the parents/caregiver and child. All those enrolled will undergo three sessions of counseling conducted by a trained nurse counselor regarding antiretroviral therapy over a two-week period.

After successful completion of the counseling process, 8 mls of blood will be drawn from each child for liver function tests, urea, blood count including hemoglobin, CD4 cell count and HIV-1 viral load.

After receiving results of the laboratory tests, children will be randomized to two groups. Those in the first group will be given a medication diary in which caregivers will record the child's daily intake of antiretroviral drugs. Those in the second group will be followed up without a diary. Children in both groups will be started on three antiretroviral drugs: zidovudine, nevirapine, and lamivudine. Caregivers will be requested to bring to the next clinic appointments drug containers for the past month's prescriptions. Those in the intervention arm will be requested to carry the medication diaries to all appointments.

Follow-up: Clinic appointments will be planned for 2 weeks after initiating antiretroviral therapy and at monthly intervals thereafter. At each visit, adherence will be monitored using self report using the pediatric adherence questionnaire. Pill counts will be performed at 3-monthly intervals. A study nurse will review the medication diary with each parent/caregiver in the intervention study arm, and address any issues raised about the diary use.

At 3,6, and 9 months after initiation of antiretroviral therapy, 8 mls of blood will be drawn from each child for liver function tests, urea, blood count including hemoglobin, CD4 cell count and HIV-1 viral load, and antiretroviral drug resistance.

In-depth interviews will be conducted with caregivers to cover a broad range of experiences.

The second two aims of this study are summarized below:

Aim 2): Define correlates of adherence measured by self report to specific components of a pediatric HAART regimen in HIV-1 infected children initiating therapy in Nairobi, Kenya.

Aim 3) Identify behavioral and social problems experienced by caregivers in relation to paediatric HAART adherence and define mechanisms to improve adherence.

ELIGIBILITY:
Inclusion Criteria:

* parents/caregivers planning to reside in Nairobi for at least one year after initiation of antiretroviral therapy
* HIV-1 infected children between ages 18 months to 12 years with symptomatic disease (WHO stage II or III) and/or CD4 <20% [where CD4 counts available]

Exclusion Criteria:

* previous use of antiretroviral drugs by the child apart from drugs taken as part of prevention of mother to child transmission of HIV
* children with end-stage AIDS including widespread disseminated malignancy, and generalized severe encephalopathy

Ages: 18 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2004-07; Primary Completion 2006-11 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
HIV-1 RNA | 9 months

SECONDARY OUTCOMES:
Follow-up CD4% and adherence | 6 months, 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Carey Farquhar, MD, MPH, Study Director — University of Washington; Dalton Wamalwa, MBChB, MPH, Principal Investigator — University of Nairobi; Grace John-Stewart, MD, PhD, Study Director — University of Washington; Dorothy Mbori-Ngacha, MBChB, MPH, Study Director — University of Nairobi; Barbra Richardson, PhD, Study Director — University of Washington; Grace Wariua, MBChB, MPH, Study Director — University of Nairobi; Julie Overbaugh, PhD, Study Director — Fred Hutchinson Cancer Center; Elizabeth Obimbo, MBChB,MPH, Study Director — University of Nairobi; Christine Gichuhi, MBChB,MMed, Study Director — University of Nairobi; Ruth Nduati, MBChB,MPH, Study Director — University of Nairobi
Locations (1):
- University of Nairobi, Nairobi, Kenya

REFERENCES:
- [Result] Farquhar C, Wamalwa D, Selig S, John-Stewart G, Mabuka J, Majiwa M, Sutton W, Haigwood N, Wariua G, Lohman-Payne B. Immune responses to measles and tetanus vaccines among Kenyan human immunodeficiency virus type 1 (HIV-1)-infected children pre- and post-highly active antiretroviral therapy and revaccination. Pediatr Infect Dis J. 2009 Apr;28(4):295-9. doi: 10.1097/INF.0b013e3181903ed3. PMID 19258919
- [Result] Wamalwa DC, Farquhar C, Obimbo EM, Selig S, Mbori-Ngacha DA, Richardson BA, Overbaugh J, Egondi T, Inwani I, John-Stewart G. Medication diaries do not improve outcomes with highly active antiretroviral therapy in Kenyan children: a randomized clinical trial. J Int AIDS Soc. 2009 Jun 24;12:8. doi: 10.1186/1758-2652-12-8. PMID 19549342
- [Result] Wamalwa DC, Farquhar C, Obimbo EM, Selig S, Mbori-Ngacha DA, Richardson BA, Overbaugh J, Emery S, Wariua G, Gichuhi C, Bosire R, John-Stewart G. Early response to highly active antiretroviral therapy in HIV-1-infected Kenyan children. J Acquir Immune Defic Syndr. 2007 Jul 1;45(3):311-7. doi: 10.1097/QAI.0b013e318042d613. PMID 17356470
- [Result] Wamalwa DC, Obimbo EM, Farquhar C, Richardson BA, Mbori-Ngacha DA, Inwani I, Benki-Nugent S, John-Stewart G. Predictors of mortality in HIV-1 infected children on antiretroviral therapy in Kenya: a prospective cohort. BMC Pediatr. 2010 May 18;10:33. doi: 10.1186/1471-2431-10-33. PMID 20482796
- [Derived] Yucha R, Litchford ML, Fish CS, Yaffe ZA, Richardson BA, Maleche-Obimbo E, John-Stewart G, Wamalwa D, Overbaugh J, Lehman DA. Higher HIV-1 Env gp120-Specific Antibody-Dependent Cellular Cytotoxicity (ADCC) Activity Is Associated with Lower Levels of Defective HIV-1 Provirus. Viruses. 2023 Oct 6;15(10):2055. doi: 10.3390/v15102055. PMID 37896832